CLINICAL TRIAL: NCT06449443
Title: Zero Echo Time MR for the Assessment of Maxillary Sinus, Bone and Soft Tissues in the Maxillary Premolar and Molar Areas
Brief Title: Zero Echo Time MR for the Assessment of Maxillary Sinus and Dental Regions
Acronym: ZTE-DENTAL
Status: Recruiting | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Guliz N. Guncu, Professor, Hacettepe University
Other Study IDs: HacettepeU21351
Record Dates: First submitted 2024-05-27; First posted 2024-06-10 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Edentulous Alveolar Ridge
Keywords: ZTE MRI; CBCT; Intraoral Scanner; Maxillary Posterior Zone; Dental Implant

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to evaluate the efficacy of zero echo time magnetic resonance imaging (ZTE MRI) as an ionizing radiation-free diagnostic method to evaluate both hard and soft tissues and maxillary sinus region before dental implants in the posterior maxillary region.

DETAILED DESCRIPTION:
Today, cone beam computed tomography (CBCT) is routinely used to evaluate the bone structure of the surgical area, to define the anatomical landmarks in the area, to detect variations, if any, and to evaluate the presence of pathologies before dental implant treatment. However, soft tissue evaluations, which are an important factor in treatment planning and the success of the treatment, cannot be performed adequately on CBCT images, and in addition, there is a significant increase in the exposure of patients to ionizing radiation. Using zero echo time magnetic resonance imaging (ZTE MRI) as a diagnostic tool that does not involve ionizing radiation in dentistry may provide a solution to this situation.

The aim of the present project is to evaluate the efficacy of ZTE MRI as an ionizing radiation-free diagnostic method to evaluate both hard and soft tissues and the maxillary sinus region before dental implants in the posterior maxillary region. For this purpose, it is planned to examine CBCT and ZTE MRI images of patients planned for dental implant treatment, to perform digital measurements with an intraoral scanner and intraoral direct measurements during surgery and to compare the results of bone and soft tissue measurements obtained.

ELIGIBILITY:
Inclusion Criteria:

* Missing teeth in the maxillary premolar and molar regions
* Cone-beam computed tomography images of the tooth-deficient area
* Do not have any systemic disease that may affect periodontal tissues (diabetes, rheumatoid arthritis, etc.)
* Over the age of 18
* Individuals who approved the informed consent form

Exclusion Criteria:

* All maxillary teeth missing
* With active periodontitis
* Under 18 years of age
* Individuals who did not approve the informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with missing teeth in the maxillary premolar and molar regions who applied to Faculty of Dentistry Department of Periodontics for dental implant treatment and who had cone beam computed tomography images for pre-surgical bone evaluation.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of maxillary sinus area with ZET-MR | Baseline-18 months
  These maxillary sinus evaluations will be conducted on both ZTE MR and CBCT images:
  1. Thickness of the sinus membrane in millimeters.
  2. Shape of thickening (dome shape or flat).
  3. Presence and characteristics of septa in the maxillary sinus. To evaluate the direction of the septum, the angle with the vertical axis will be measured; then the direction of the septum will be classified as vertical (<30°), oblique (between 30° and 60°), and horizontal (between 60° and 90°). In terms of morphology, if the septum extends from one sinus wall to the opposite sinus wall, it will be classified as 'complete'; if it does not reach the opposite wall, it will be considered 'partial'.
  4. Presence and variations of the posterior superior alveolar artery (intraosseous or below the membrane or on the outer cortex of the lateral sinus wall)
  5. Diameter of the artery and distances to the sinus floor and alveolar crest in millimeters.
  6. Thickness of the lateral sinus wall in milimeters.
Evaluation of alveolar bone dimensions in maxillary premolar and molar areas with ZET-MR, CBCT and directly | Baseline-18 months
  These assessments will be conducted on both preoperative CBCT and zero echo time MR images, as well as directly during surgery using a caliper.
  * Repeated bone thickness measurements at 1, 3, 5, 7, and 9 mm points relative to the crest top
  * The bone height from the crest top to the sinus floor at 5 mm mesiodistally from the last tooth
Evaluation of soft tissue for dental implant planning Evaluation of gingival tissue dimensions in maxillary premolar and molar areas with ZET-MR and directly during surgery | Baseline -18 months
  Gingival thickness measurements will be performed at 2, 4, and 6 mm apically from the alveolar crest through to apical area with three different methods:
  1. ZET-MR images in milimeters.
  2. Intraoral scanner images overlapped with CBCT data in milimeters.
  3. Clinically during dental implant surgery with a periodontal probe after local anesthesia in milimeters.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Department of Periodontology, Faculty of Dentistry, Hacettepe University,, Ankara
  - Hacettepe University Faculty of Medicine, Ankara